CLINICAL TRIAL: NCT00592397
Title: Prestudy: Lifestyle and Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); FUGE Mid-Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REK 4.2005.2187; 13714 (Other: NSD)
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Diabetes Mellitus; Cardiovascular Diseases
Keywords: Dietary Intervention; Nutrigenomics; Diet, Carbohydrate-Restricted; Gene Expression; Gene Expression Profiling; Oligonucleotide Array Sequence Analysis; Biological Markers; Food; Obesity; Blood; Subcutaneous Fat, Abdominal
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All participants underwent the same dietary intervention
  Interventions: Other: Balanced macronutrient diet intervention

INTERVENTIONS:
Other: Balanced macronutrient diet intervention — Isocaloric dietary changes from typically Western diet to balanced macronutrient composition.
  Other Names: Microarray study of diet intervention

SUMMARY:
The purpose of this pilot study is to optimize conditions for a planned human intervention study focusing on how diet predispose for, and influence, lifestyle disease development and its consequence in cardiovascular disease development.

DETAILED DESCRIPTION:
Common for many of the risk factors of lifestyle diseases is that they are induced by improper diet. Recent research has shown that especially total amount and composition of the macro nutrients, protein, carbohydrate and fats, is important.

A time course experiment has been performed where 5 subjects underwent a diet intervention for four weeks with a controlled, balanced macro nutrient energy content of every meal. The sampling time points were 0, 1, 2, 7, 14 and 28 days. The goals were to determine optimal length of intervention with stabilization of gene expression to occur and compare blood and subcutaneous abdominal fat tissue as source of biological material for RNA for DNA microarray analysis. Microarray analysis were performed on 3 of the 5 subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy males, BMI>30

Exclusion Criteria:

* known chronic disease or in need of any medical treatment

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Changes in microarray gene expression profiles in blood and subcutaneous abdominal fat tissue from healthy obese men, as a consequence of changes in dietary macro nutrient composition. | Four weeks

SECONDARY OUTCOMES:
Time to stabilization of gene expression changes due to dietary intervention. | 0, 1, 2, 7, 14 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Berit Johansen, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Mid-Norway, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brattbakk HR, Arbo I, Aagaard S, Lindseth I, de Soysa AK, Langaas M, Kulseng B, Lindberg F, Johansen B. Balanced caloric macronutrient composition downregulates immunological gene expression in human blood cells-adipose tissue diverges. OMICS. 2013 Jan;17(1):41-52. doi: 10.1089/omi.2010.0124. Epub 2011 Jun 16. PMID 21679058